CLINICAL TRIAL: NCT05683327
Title: The Effect of Oral Hyaluronic Acid (UltraHA®) on the Knee Function: A Randomized-Blind, Placebo-Controlled Study
Brief Title: The Effect of Oral Hyaluronic Acid (UltraHA®) on the Knee Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthomedico Inc. (Other)
Collaborators: BLOOMAGE BIOTECHNOLOGY CORPORATION LIMITED (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06793-0003-0E
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-01

CONDITIONS: Healthy Japanese Subjects
Keywords: Hyaluronic Acid; Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hyaluronic Acid 150 mg (Active Comparator): Take 150 mg/day of hyaluronic acid.
  Interventions: Dietary Supplement: UltraHA® 75 mg/capsule
- Hyaluronic Acid 80 mg (Active Comparator): Take 80 mg/day of hyaluronic acid.
  Interventions: Dietary Supplement: UltraHA® 40 mg/capsule
- Placebo (Placebo Comparator): Take 0 mg/day of hyaluronic acid.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: UltraHA® 75 mg/capsule — Take 2 capsules per day at any time.
  Arms: Hyaluronic Acid 150 mg
Dietary Supplement: UltraHA® 40 mg/capsule — Take 2 capsules per day at any time.
  Arms: Hyaluronic Acid 80 mg
Dietary Supplement: Placebo — Take 2 capsules per day at any time.
  Arms: Placebo

SUMMARY:
This clinical trial aims to clarify the effect of UltraHA® on knee joint conditions.

DETAILED DESCRIPTION:
In this study, the investigators will evaluate the knee condition before and after the intervention. The groups to be compared are two different doses of UltraHA® and a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese
2. Men or women
3. Adults
4. Healthy subjects
5. Subjects whose skin viscoelasticity is relatively low at screening (before consumption)
6. Subjects whose BMI are 23 kg/m^2 or more and less than 30 kg/m^2
7. Subjects who are judged in the Kellgren-Lawrence grade (KL grade) as either 0 or 1 in X-ray
8. Subjects whose WOMAC score is relatively high

Exclusion Criteria:

1. Subjects who are undergoing medical treatment or have a medical history of malignant tumor, heart failure, and myocardial infarction
2. Subjects who have a pacemaker or an implantable cardioverter defibrillator (ICD)
3. Subjects currently undergoing treatment for any of the following chronic diseases: cardiac arrhythmia, liver disorder, kidney disorder, cerebrovascular disorder, rheumatism, diabetes mellitus, dyslipidemia, hypertension, or any other chronic diseases
4. Subjects who use or take "Foods for Specified Health Uses," or "Foods with Functional Claims" in daily
5. Subjects who consciously consume foods that contribute to knee joint improvements, such as collagen and chondroitin sulfate
6. Subjects who are currently taking medications (including herbal medicines) and supplements
7. Subjects who are allergic to medications and/or the test-food-related products (particularly alcohol)
8. Subjects who are pregnant, lactating, or planning to become pregnant during this trial
9. Subjects who suffer from COVID-19
10. Subjects who have been enrolled in other clinical trials within the last 28 days before the agreement to participate in this trial or plan to participate another trial during this trial
11. Subjects who are judged as ineligible to participate in this study by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scores at Week 12 | Week 12
  The WOMAC contains 24 questions, including pain for 5 questions, stiffness for 2 questions, and physical function for 17 questions, answered on a range of 0 (mildest) to 4 (most severe). The sum of responses is evaluated as the WOMAC scores.

SECONDARY OUTCOMES:
Each WOMAC subscale score at Week 12 | Week 12
  The WOMAC contains 24 questions, including pain for 5 questions, stiffness for 2 questions, and physical function for 17 questions, answered on a range of 0 (mildest) to 4 (most severe). The sum of each subscale response is evaluated as the WOMAC subscale score.
Subjective symptoms at Week 12 | Week 12
  Assess knee pain, stiffness, discomfort, and health using visual analogue scale. There is a 100 mm straight line with the best and worst degree of sensation indicated at both ends, and the current degree of sensation is marked on the line with the best imaginable state being 0 and the worst state being 100.

CONTACTS AND LOCATIONS:
Overall Officials: Tsuyoshi Takara, MD, Study Chair — Medical Corporation Seishinkai, Takara Clinic
Locations (2):
- Japan (2):
  - Nerima Medical Association Minami-machi Clinic, Nerima-ku, Tokyo
  - Medical Corporation Seishinkai, Takara Clinic, Shinagawa-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No
Data sharing will be discussed among the research affiliates after the study is completed.